CLINICAL TRIAL: NCT00808054
Title: Evaluation of Analgesia With the Use of Eutectic Mixture of Local Anesthetics (Lidocaine and Prilocaine) and Oral Solution of Glucose to 25% in Preterm Neonates During Arterial Puncture and / or the Installation of Percutaneous Catheter
Brief Title: Evaluation of Analgesia With EMLA and Glucose Oral Solution
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Renato Santiago Gomez, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CAAE0049028720308
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Pain
Keywords: Pain; preterm neonate; pain assessment; EMLA; oral glucose
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glucose and EMLA (Experimental): Received glucose oral and topical EMLA
  Interventions: Drug: EMLA
- Glucose and placebo (Experimental): Received glucose and no EMLA
  Interventions: Drug: EMLA
- Oral placebo and EMLA (Experimental): Received oral placebo and EMLA
  Interventions: Drug: EMLA

INTERVENTIONS:
Drug: EMLA — 0.5g topical EMLA
  Other Names: Lidocaine and prilocaine cream

SUMMARY:
In this randomized controlled study the investigators intended to compare analgesic effects of EMLA and/or oral glucose in 60 preterm neonate during arterial function and PICC installation.

DETAILED DESCRIPTION:
It is a randomised controlled clinical trial, double blinded, with the purpose to compare the use of eutectic mixture of local anesthetics (lidocaine and prilocaine) and/or the oral solution of glucose 25% in the prevention and treatment of pain in preterm neonates with gestational between 28-37 weeks old.

The pain evaluation will be done using NIPS scale, and also physiologic variables (HR, MAP, oxygen saturation level and crie) during two painful procedures performed in the neonatal intensive care units:arterial puncture (n=30) and peripherally inserted central catheters (n=30). All procedures will have clinical indication and will not be implemented by the researcher.The newborns will be randomized into three groups: A (EMLA and glucose; n=20),B (EMLA AND placebo; n=20) and C (anesthetic cream placebo and oral glucose; n=20).

All newborns will be subjected to some kind of therapeutic intervention, the objective of this study is validate the application of control measures and treatment of pain for these two procedures that cause mild and moderate pain.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age greater than or equal to 28 weeks and less than 37 weeks
2. Admission in the neonatal intensive care unit of the hospital Julia Kubtischek
3. Clinical indication of collection of blood through arterial puncture or peripherally inserted central catheter
4. Neonate in the first week of life (first to seventh day of life);
5. Informed consent have to be obtained by parents or guardians.

Exclusion Criteria:

1. Newborn with broken skin at cream application site;
2. Use of sedation or analgesia in the last 72 hours;
3. Diagnosis of necrotizing enterocolitis;
4. Anemia
5. Metabolic acidosis
6. Methaemoglobinaemia
7. Treatment with agents to induce methemoglobinemia
8. Mechanical ventilation in patients using opioids
9. Clinical diagnosis of neuromuscular dysfunction
10. Any contraindication to suction
11. Urgent procedures

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Compare analgesic efficacy of EMLA versus oral glucose | From the first to seven day of life

SECONDARY OUTCOMES:
Evaluate analgesic synergism of EMLA versus oral glucose | First to seven day of life

CONTACTS AND LOCATIONS:
Overall Officials: Yerkes Pereira Silva, PhD, Principal Investigator — Federal University of Minas gerai
Locations (1):
- Department of Neonatology of Julia Kubitschek Hospital, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Lehr VT, Taddio A. Topical anesthesia in neonates: clinical practices and practical considerations. Semin Perinatol. 2007 Oct;31(5):323-9. doi: 10.1053/j.semperi.2007.07.008. PMID 17905188
- [Background] Taddio A, Ohlsson A, Einarson TR, Stevens B, Koren G. A systematic review of lidocaine-prilocaine cream (EMLA) in the treatment of acute pain in neonates. Pediatrics. 1998 Feb;101(2):E1. doi: 10.1542/peds.101.2.e1. PMID 9445511
- [Background] Deshmukh LS, Udani RH. Analgesic effect of oral glucose in preterm infants during venipuncture--a double-blind, randomized, controlled trial. J Trop Pediatr. 2002 Jun;48(3):138-41. doi: 10.1093/tropej/48.3.138. PMID 12164596